CLINICAL TRIAL: NCT01956812
Title: An International, Multi-Center, Double-Blind, Randomized, Phase III Trial of 90Y-Clivatuzumab Tetraxetan Plus Low-Dose Gemcitabine Versus Placebo Plus Low-Dose Gemcitabine in Patients With Metastatic (Stage IV) Pancreatic Adenocarcinoma Who Received at Least Two Prior Treatments (PANCRIT-1)
Brief Title: Phase 3 Trial of 90Y-Clivatuzumab Tetraxetan & Gemcitabine vs Placebo & Gemcitabine in Metastatic Pancreatic Cancer
Acronym: PANCRIT®-1
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The DSMB conducted an interim analysis on overall survival, which showed that the treatment arm did not demonstrate a sufficient improvement in OS vs. placebo.
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IMMU-107-04
Record Dates: First submitted 2013-09-26; First posted 2013-10-08 (Estimated); Last update posted 2021-08-16 (Actual); Status verified 2020-03

CONDITIONS: Metastatic Pancreatic Cancer; Pancreatic Cancer
Keywords: clivatuzumab tetraxetan; 90Y-clivatuzumab tetraxetan; IMMU-107
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Saline Solution; Gemcitabine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A IMMU-107 and gemcitabine (Experimental): IMMU-107 and low dose gemcitabine
  Interventions: Drug: IMMU-107; Drug: Gemcitabine
- Arm B Placebo and low dose gemcitabine (Active Comparator): Placebo and low dose gemcitabine
  Interventions: Drug: placebo; Drug: Gemcitabine

INTERVENTIONS:
Drug: IMMU-107 — Arm A: gemcitabine 200 mg/m2 administered weekly x 4 and IMMU-107 administered weekly x 3 for multiple cycles
  Other Names: 90Y-clivatuzumab tetraxetan
  Arms: Arm A IMMU-107 and gemcitabine
Drug: placebo — placebo weekly x 3 and gemcitabine 200 mg/m2 weekly x 4 for multiple cycles
  Other Names: normal saline
  Arms: Arm B Placebo and low dose gemcitabine
Drug: Gemcitabine — Gemcitabine, 200 mg/m2, given weekly x 4 in both arms
  Other Names: gemcitabine 200 mg/m2

SUMMARY:
The is a double-blind, randomized phase 3 study of 90Y-clivatuzumab tetraxetan with low-dose gemcitabine, versus placebo and low-dose gemcitabine in metastatic pancreatic cancer patients who have progressed on at least 2 prior therapies for metastatic cancer (1 of which was a gemcitabine-containing regimen).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the pancreas
* Metastatic disease
* Received at least two prior systemic cytotoxic chemotherapy regimens for unresectable, locally advanced or metastatic disease.
* At least one of the prior systemic cytotoxic chemotherapy regimens for unresectable, locally advanced or metastatic disease must have contained gemcitabine and have met the following criteria:
* Completed at least one cycle of the treatment
* Received gemcitabine administered at a minimum dose of 800 mg/m2 per week in the first cycle of treatment
* Progressed while receiving this gemcitabine regimen or within 3 months of completing gemcitabine
* Progression was documented,
* Preferentially radiologically by tumor growth or new lesions, or by
* Clear symptomatic deterioration supported by at least two of the following clinical criteria: ≥ 10% worsening in KPS or ≥ 1 worsening in ECOG; increasing weakness or fatigue; progressive weight loss; new/worsening pain requiring increased pain medication; new/worsening jaundice, nausea, or vomiting; new/worsening ascites or pleural effusions; other physical or laboratory findings consistent with disease progression.
* KPS >/= 70
* Adequate bone marrow function
* Adequate hepatic function
* Adequate renal function

Exclusion Criteria:

* CNS metastatic disease
* Bulky disease (any single mass >10 cm).

  ->Grade 2 nausea or vomiting, and/or signs of intestinal obstruction.
* Prior external beam irradiation to a field that includes more than 30% of the red bone marrow.
* Patients with clinically significant severe cardiorespiratory disease.

Please consult with the clinical trial site for the full detailed list of specific inclusion/exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 334 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
overall survival | 24 months

SECONDARY OUTCOMES:
Overall survival | 3, 6 and 12 months
Objective tumor response | 24 months
Progression free survival | 24 months
Clinical benefit | 24 months
  quality of life will be assessed over 24 months using the FACT-hepatopancreatic form

CONTACTS AND LOCATIONS:
Overall Officials: William Wegener, MD, PhD, Study Chair — Gilead Sciences
Locations (64):
- United States (42):
  - Banner MD Anderson, Gilbert, Arizona
  - City of Hope National Medical Center, Duarte, California
  - Pacific Shores Medical Group, Long Beach, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Whittingham Cancer Center, Norwalk, Connecticut
  - Michael and Dianne Bienes Comprehensive Cancer Center - Holy Cross Hospital, Fort Lauderdale, Florida
  - Baptist Cancer Institute, Jacksonville, Florida
  - Cancer Specialists of North Florida, Jacksonville, Florida
  - Mountain States Tumor Institute at St. Luke's Regional Medical Center, Boise, Idaho
  - Illinois Cancer Specialists, Arlington Heights, Illinois
  - Indiana University Health Goshen Center for Cancer Care, Goshen, Indiana
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Ashland-Bellefonte Cancer Center, Ashland, Kentucky
  - University of Maryland Medical Center, Baltimore, Maryland
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Oncology Hematology West P.C. dba Nebraska Cancer Specialists, Omaha, Nebraska
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - New York Presbyterian Hospital/Weill Cornell Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - University of North Carolina Hospitals, Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - The Ohio State University - Comprehensive Cancer Center, Columbus, Ohio
  - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - The Pennsylvania State University (Penn State) Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania Abramson Cancer Center, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center/Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Center for Biomedical Research, Knoxville, Tennessee
  - University of Tennessee Medical Center, Cancer Institute, Knoxville, Tennessee
  - Mary Crowley Medical Research Center, Dallas, Texas
  - Oncology Consultants, Houston, Texas
  - Texas Oncology - McAllen, McAllen, Texas
  - Texas Oncology - Tyler, Tyler, Texas
  - Virginia Oncology Associates, Norfolk, Virginia
  - University of Washington, Seattle, Washington
  - Virginia Mason Medical Center, Seattle, Washington
- Austria (2):
  - Krankenhaus der Elisabethinen Linz, Linz
  - Medical University Vienna, Vienna
- University Hospital Leuven, Leuven, Belgium
- Canada (2):
  - Cancer Care Manitoba, Winnepeg, Manitoba
  - Centre Hospitalier Université de Sherbrooke, Sherbrooke, Quebec
- France (7):
  - ICO René Gauducheau, Nantes, Cedex 1
  - Institut Paoli-Calmettes, Marseille, Cedex 9
  - Institut Bergonie, Bordeaux, Cedex
  - Centre Léon Bérard Cancerologie Medicale, Lyon
  - Institut Paoli-Calmettes, Marseille
  - CRLC Val D'Aurelle, Montpellier
  - Hopital Cochin, Paris
- Israel (2):
  - Soroka Medical Center, Beersheba
  - Rambam Medical Center, Haifa
- Centrum Onkologii Instytut im. M. Sklodowskiej-Curie - Warszawa, Warsaw, Poland
- Spain (7):
  - Hospital Sant Joan de Reu, Reus, Tarragona
  - Hospital Vall D'Hebrón, Barcelona
  - Hospital Universitario Gregorio Marañón, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario La Paz, Madrid
  - Centro Integral Oncologico Clara Campal, Madrid
  - Hospital Miguel Servet, Zaragoza

REFERENCES:
- [Background] Ocean AJ, Pennington KL, Guarino MJ, Sheikh A, Bekaii-Saab T, Serafini AN, Lee D, Sung MW, Gulec SA, Goldsmith SJ, Manzone T, Holt M, O'Neil BH, Hall N, Montero AJ, Kauh J, Gold DV, Horne H, Wegener WA, Goldenberg DM. Fractionated radioimmunotherapy with (90) Y-clivatuzumab tetraxetan and low-dose gemcitabine is active in advanced pancreatic cancer: A phase 1 trial. Cancer. 2012 Nov 15;118(22):5497-506. doi: 10.1002/cncr.27592. Epub 2012 May 8. PMID 22569804
- [Background] Gulec SA, Cohen SJ, Pennington KL, Zuckier LS, Hauke RJ, Horne H, Wegener WA, Teoh N, Gold DV, Sharkey RM, Goldenberg DM. Treatment of advanced pancreatic carcinoma with 90Y-Clivatuzumab Tetraxetan: a phase I single-dose escalation trial. Clin Cancer Res. 2011 Jun 15;17(12):4091-100. doi: 10.1158/1078-0432.CCR-10-2579. Epub 2011 Apr 28. PMID 21527562
- [Background] Sharkey RM, Karacay H, Govindan SV, Goldenberg DM. Combination radioimmunotherapy and chemoimmunotherapy involving different or the same targets improves therapy of human pancreatic carcinoma xenograft models. Mol Cancer Ther. 2011 Jun;10(6):1072-81. doi: 10.1158/1535-7163.MCT-11-0115. Epub 2011 Apr 5. PMID 21467164
- [Background] Tokh M, Bathini V, Saif MW. First-line treatment of metastatic pancreatic cancer. JOP. 2012 Mar 10;13(2):159-62. PMID 22406590
- [Background] Gold DV, Newsome G, Liu D, Goldenberg DM. Mapping PAM4 (clivatuzumab), a monoclonal antibody in clinical trials for early detection and therapy of pancreatic ductal adenocarcinoma, to MUC5AC mucin. Mol Cancer. 2013 Nov 20;12(1):143. doi: 10.1186/1476-4598-12-143. PMID 24257318
- [Background] Gold DV, Gaedcke J, Ghadimi BM, Goggins M, Hruban RH, Liu M, Newsome G, Goldenberg DM. PAM4 enzyme immunoassay alone and in combination with CA 19-9 for the detection of pancreatic adenocarcinoma. Cancer. 2013 Feb 1;119(3):522-8. doi: 10.1002/cncr.27762. Epub 2012 Aug 16. PMID 22898932
- [Background] Gold DV, Goggins M, Modrak DE, Newsome G, Liu M, Shi C, Hruban RH, Goldenberg DM. Detection of early-stage pancreatic adenocarcinoma. Cancer Epidemiol Biomarkers Prev. 2010 Nov;19(11):2786-94. doi: 10.1158/1055-9965.EPI-10-0667. Epub 2010 Sep 1. PMID 20810605
- [Background] Gold DV, Goldenberg DM, Karacay H, Rossi EA, Chang CH, Cardillo TM, McBride WJ, Sharkey RM. A novel bispecific, trivalent antibody construct for targeting pancreatic carcinoma. Cancer Res. 2008 Jun 15;68(12):4819-26. doi: 10.1158/0008-5472.CAN-08-0232. PMID 18559529
- [Background] Gold DV, Karanjawala Z, Modrak DE, Goldenberg DM, Hruban RH. PAM4-reactive MUC1 is a biomarker for early pancreatic adenocarcinoma. Clin Cancer Res. 2007 Dec 15;13(24):7380-7. doi: 10.1158/1078-0432.CCR-07-1488. PMID 18094420
- [Background] Gold DV, Modrak DE, Ying Z, Cardillo TM, Sharkey RM, Goldenberg DM. New MUC1 serum immunoassay differentiates pancreatic cancer from pancreatitis. J Clin Oncol. 2006 Jan 10;24(2):252-8. doi: 10.1200/JCO.2005.02.8282. Epub 2005 Dec 12. PMID 16344318
- [Background] Gold DV, Modrak DE, Schutsky K, Cardillo TM. Combined 90Yttrium-DOTA-labeled PAM4 antibody radioimmunotherapy and gemcitabine radiosensitization for the treatment of a human pancreatic cancer xenograft. Int J Cancer. 2004 Apr 20;109(4):618-26. doi: 10.1002/ijc.20004. PMID 14991585
- [Background] Gold DV, Schutsky K, Modrak D, Cardillo TM. Low-dose radioimmunotherapy ((90)Y-PAM4) combined with gemcitabine for the treatment of experimental pancreatic cancer. Clin Cancer Res. 2003 Sep 1;9(10 Pt 2):3929S-37S. PMID 14506191
- [Background] Cardillo TM, Blumenthal R, Ying Z, Gold DV. Combined gemcitabine and radioimmunotherapy for the treatment of pancreatic cancer. Int J Cancer. 2002 Jan 20;97(3):386-92. doi: 10.1002/ijc.1613. PMID 11774294
- [Background] Cardillo TM, Ying Z, Gold DV. Therapeutic advantage of (90)yttrium- versus (131)iodine-labeled PAM4 antibody in experimental pancreatic cancer. Clin Cancer Res. 2001 Oct;7(10):3186-92. PMID 11595713
- [Background] Gold DV, Cardillo T, Goldenberg DM, Sharkey RM. Localization of pancreatic cancer with radiolabeled monoclonal antibody PAM4. Crit Rev Oncol Hematol. 2001 Jul-Aug;39(1-2):147-54. doi: 10.1016/s1040-8428(01)00114-7. PMID 11418312
- [Background] Gold DV, Cardillo T, Vardi Y, Blumenthal R. Radioimmunotherapy of experimental pancreatic cancer with 131I-labeled monoclonal antibody PAM4. Int J Cancer. 1997 May 16;71(4):660-7. doi: 10.1002/(sici)1097-0215(19970516)71:43.0.co;2-e. PMID 9178823
- [Background] Mariani G, Molea N, Bacciardi D, Boggi U, Fornaciari G, Campani D, Salvadori PA, Giulianotti PC, Mosca F, Gold DV, et al. Initial tumor targeting, biodistribution, and pharmacokinetic evaluation of the monoclonal antibody PAM4 in patients with pancreatic cancer. Cancer Res. 1995 Dec 1;55(23 Suppl):5911s-5915s. PMID 7493369
- [Background] Alisauskus R, Wong GY, Gold DV. Initial studies of monoclonal antibody PAM4 targeting to xenografted orthotopic pancreatic cancer. Cancer Res. 1995 Dec 1;55(23 Suppl):5743s-5748s. PMID 7493339
- [Background] Gold DV, Lew K, Maliniak R, Hernandez M, Cardillo T. Characterization of monoclonal antibody PAM4 reactive with a pancreatic cancer mucin. Int J Cancer. 1994 Apr 15;57(2):204-10. doi: 10.1002/ijc.2910570213. PMID 7512537